CLINICAL TRIAL: NCT06495814
Title: Characterization and Mechanism Research of the Pre-disease State of Obese Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fengmei Lian (Other)
Responsible Party: Sponsor-Investigator, Fengmei Lian, Researcher, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obese type 2 diabetes mellitus
Record Dates: First submitted 2024-07-02; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Obese Impaired Glucose Tolerance; Newly Diagnosed Obese Type 2 Diabetic Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cross sectional group of newly diagnosed obese type 2 diabetes mellitus (No Intervention): No intervention conducted
- Cross section group of healthy individuals (No Intervention): No intervention conducted
- Intervention group of high-risk obese impaired glucose tolerance (Experimental): General lifestyle intervention+1/bag of Jinlida granules, 3 times/day, taken with hot water.
  Interventions: Drug: 1/bag of Jinlida granules, 3 times/day, taken with hot water.
- Observation group of high-risk obese impaired glucose tolerance (No Intervention): General lifestyle intervention
- Observation group of low-risk obese impaired glucose tolerance (No Intervention): General lifestyle intervention
- Cross sectional group and observation group of obese impaired glucose tolerance (No Intervention): General lifestyle intervention

INTERVENTIONS:
Drug: 1/bag of Jinlida granules, 3 times/day, taken with hot water. — All observation and intervention groups received lifestyle interventions, with only the intervention group of high-risk obese impaired glucose tolerance receiving intervention with Jinlida granules.
  Other Names: General lifestyle intervention
  Arms: Intervention group of high-risk obese impaired glucose tolerance

SUMMARY:
Establish a comprehensive evaluation system for the progression of obese impaired glucose tolerance (IGT) to type 2 diabetes mellitus (T2DM) through cross-sectional studies; Constructing and validating a T2DM risk prediction model for obese IGT population through observational research; Through open-label clinical research, we applied Jinlida granules to intervene in high-risk obese IGT population and clarify its protective effect on this population.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for obese IGT population:

* Age range from 18 to 65 years old, including both ends;

  * Meet the waist circumference cut-off point for central obesity diagnosis specified in the "Guidelines for Primary Diagnosis and Treatment of Obesity (2019)";

    * Meet the IGT diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Type 2 diabetes (2020 Edition);

      * Voluntarily participate in this study and sign an informed consent form.

Inclusion criteria for newly diagnosed obese T2DM population:

① Age range from 18 to 65 years old, including both ends;

② Meet the waist circumference cut-off point for central obesity diagnosis specified in the "Guidelines for Primary Diagnosis and Treatment of Obesity (2019)";

③ Conform to the T2DM diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Type 2 diabetes (2020 Edition), and the course of disease is less than 3 months;

* Voluntarily participate in this study and sign an informed consent form.

Inclusion criteria for healthy individuals:

* Age range from 18 to 65 years old, including both ends;

  * Meets the diagnostic criteria for healthy individuals set by WHO;

    * Voluntarily sign an informed consent form.

Inclusion criteria for IGT for high and low-risk obesity:

* Age range from 18 to 65 years old, including both ends;

  * Meet the waist circumference cut-off point for central obesity diagnosis specified in the "Guidelines for Primary Diagnosis and Treatment of Obesity (2019)";

    * Meet the IGT diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Type 2 diabetes (2020 Edition);

      * After screening the risk prediction model constructed in this study, it belongs to the high-risk and low-risk populations with abnormal glucose tolerance;

        * Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

Exclusion criteria for obese IGT patients:

* The population who have been continuously using hypoglycemic drugs within the past three months;

  * Type 1 diabetes and type 2 diabetes (T2DM), pregnancy diabetes, secondary diabetes and other special types of diabetes;

    * Hyperthyroidism or hypothyroidism caused by endocrine disorders, with poor disease control;

      * Difficult to control hypertension/hypotension: systolic blood pressure ≥ 200mmHg or diastolic blood pressure ≥ 110mmHg; Or systolic blood pressure ≤ 90mmHg or diastolic blood pressure ≤ 60mmHg;

        * When screening, patients with various acute infections, or those accompanied by severe infections, severe anemia, or neutropenia;

          * Accompanied by other major diseases, such as active or untreated malignant tumors, or clinical remission of malignant tumors for less than 5 years;

            * Organic heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, with NYHA heart function grading>Grade III;

              ⑧ The patient has suffered from any of the following diseases within the past 6 months: coronary intervention (such as CABG or PTCA), stroke (including ischemic and hemorrhagic stroke);

              ⑨ Severe liver and kidney dysfunction (ALT greater than 3 times the upper normal limit, creatinine greater than 132 μ mol/l);

              ⑩ Fasting TG>5.6mmol/L;

              ⑪ Pregnant and lactating women, as well as women of childbearing age who have not taken effective contraceptive measures;

              ⑫ Participating in any other clinical trials/researchers;

              ⑬ Patients with a history of alcoholism or long-term drug abuse;

              ⑭ Individuals with a history of mental illness are unable to cooperate with the researchers;

              ⑮ For any other reason, the researcher considers it unsuitable to participate in this study.

Exclusion criteria for newly diagnosed obese T2DM patients:

* Type 1 diabetes, gestational diabetes, secondary diabetes and other special types of diabetes;

  * The population who have been continuously using hypoglycemic drugs within the past three months;

    * Patients with complications of diabetes;
    * Hyperthyroidism or hypothyroidism caused by endocrine disorders, with poor disease control;

      * Difficult to control hypertension/hypotension: systolic blood pressure ≥ 200mmHg or diastolic blood pressure ≥ 110mmHg; Or systolic blood pressure ≤ 90mmHg or diastolic blood pressure ≤ 60mmHg;

        * When screening, patients with various acute infections, or those accompanied by severe infections, severe anemia, or neutropenia;

          * Accompanied by other major diseases, such as active or untreated malignant tumors, or clinical remission of malignant tumors for less than 5 years;

            ⑦ Organic heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, with NYHA heart function grading>Grade III;

            ⑧ The patient has suffered from any of the following diseases within the past 6 months: coronary intervention (such as CABG or PTCA), stroke (including ischemic and hemorrhagic stroke);

            ⑨ Severe liver and kidney dysfunction (ALT greater than 3 times the upper normal limit, creatinine greater than 132 μ mol/l);

            ⑩ Fasting TG>5.6mmol/L;
            * Pregnant and lactating women, as well as women of childbearing age who have not taken effective contraceptive measures;

              * Patients with a history of alcoholism or long-term drug abuse;

                * Individuals with a history of mental illness are unable to cooperate with the researchers;

                  * Participating in any other clinical trials/researchers;

                    ⑮ For any other reason, the researcher considers it unsuitable to participate in this study.

Exclusion criteria for healthy individuals:

* Any history of chronic diseases of various systems that have been previously diagnosed, such as obesity, endocrine and metabolic diseases, hematopoietic system diseases, respiratory system diseases, cardiovascular system diseases, malignant tumors, liver and kidney dysfunction, etc;

  * When screening, patients with various acute infections, or those accompanied by severe infections, severe anemia, or neutropenia;

    * Patients with a history of alcoholism or long-term drug abuse;

      * Pregnant or lactating women;

        * Individuals with a history of mental illness who cannot cooperate with the research process;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of diabetes | Both the observation group and the intervention group were followed up for 12 months, once a month.
  During the follow-up period, when the subjects measured abnormal fasting blood glucose, venous blood was collected and OGTT was measured. Subjects who were diagnosed with type 2 diabetes according to the OGTT results and who were still diagnosed with type 2 diabetes by OGTT one week later were defined as the occurrence of diabetes.

IPD SHARING:
Plan to Share IPD: No